CLINICAL TRIAL: NCT05173740
Title: The ROCK Trial. A Multidisciplinary Rehabilitation Intervention Targeted Return-to-work in Sudden Out-of-hospital Cardiac Arrest Survivors A Pragmatic Randomised Controlled Trial
Brief Title: Rehabilitation for Survivors of Out-of-hospital Cardiac Arrest
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Jan Christensen, Senior Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20049654
Record Dates: First submitted 2021-11-27; First posted 2021-12-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest; Heart Arrest; Cardiopulmonary Resuscitation; Return to Work; Return-to-work; Rehabilitation; Recovery of Function; Cardiac Rehabilitation
Keywords: Labour marked; Cardiac arrest; Heart Arrest; Cardiopulmonary Resuscitation; Return to work; Return-to-work; Back to Work; Rehabilitation; Recovery of Function; Cardiac Rehabilitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Before data extraction and data analysis all data will be anonymized, and group allocation will be blinded as (group X and Y).
  Participants will be randomly assigned to either the intervention or the usual care group using a computer random generator, with a 1:1 allocation. The randomisation will be conducted by a blinded investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individually tailored rehabilitation intervention + usual care (Experimental): A comprehensive neurocognitive assessment and a thorough individual assessment of rehabilitation needs will be conducted to inform the individually tailored intervention plan. Core intervention elements are: 1) comprehensive assessment of individual rehabilitation needs including neuropsychology tests in order to make a individually tailored intervention plan coordinated with the multidisciplinary rehabilitation team, 2) providing strategies to lessen impact for the individual cognitive impairment, 3) educating survivors and relatives about the impact of a cardiac arrest and consequences on daily life, 4) work preparation, including establishment of routines and opportunities to practice work skills and 5) collaboration with the local municipality's job centre and employers to plan, support and monitor graded RTW, 6) short term therapy by psychologist dealing with thoughts and behaviour in relation to cardiac arrest.
  Interventions: Other: Individually tailored rehabilitation intervention
- Usual care (Active Comparator): All participants including those allocated to the usual care group will be seen by an occupational therapist if their MoCA screening score ≤26. Furthermore, if considered relevant by the discharging unit, survivors are referred for rehabilitation provided and delivered in the local municipality where the participant is resident. The content of the rehabilitation will typically be based on the content of the rehabilitation plan from the discharging hospital unit and an individual assessment of the survivors' expressed needs, within the local municipality where the participant is resident.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Individually tailored rehabilitation intervention — Individually tailored rehabilitation intervention
  Arms: Individually tailored rehabilitation intervention + usual care
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
This study is a parallel group multicentre investigator-initiated clinical randomised controlled superiority trial that will include a total of 214 survivors of OHCA.

Participants will to be randomized with a 1:1 allocation ratio to either a intervention consisting of a comprehensive initiated tailored rehabilitation intervention focusing on supporting RTW plus usual care compared to usual care alone.

DETAILED DESCRIPTION:
The ROCK trial is a two-arm multicentre investigator-initiated clinical randomised controlled superiority trial evaluating the effectiveness of a comprehensive individually tailored rehabilitation intervention focusing on supporting labour marked participation of survivors of out-of-hospital cardiac arrest compared to usual care, with primary endpoint measured after 12 months follow-up.

The overall aim of the ROCK trial is to evaluate the effectiveness of a comprehensive individually tailored multidisciplinary rehabilitation intervention for survivors of OHCA on RTW compared to usual care. The investigators hypothesize that the intervention will result in a higher-level labour marked attachment one year after hospital discharge in addition to increased health-related quality of life.

A full statistical analysis plan describing all details have been developed. In short, data from the national register on social transfer payments (DREAM database) will form the basis for the primary outcome. The primary outcome is labour market participation, defined as the proportion of employment vs. on social transfer payment, and the primary end point will be collected 12 months after hospital discharge.

ELIGIBILITY:
Inclusion criteria:

* All adult survivors with first time out-of-hospital cardiac arrest
* Discharged from the Hospitals will be assessed eligible for inclusion

Exclusion criteria:

* Survivors who prior to the cardiac arrest were not part of the labour force with at least two years until they are qualified to receive retirement state pensions
* Patients that cannot understand and fulfil the study surveys (in Danish)
* Patients with short witnessed cardiac arrests with return of spontaneous circulation estimated less than 4 minutes and immediate awakening without ICU treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Labour market participation using data from the DREAM database | 12-months after hospital discharge
  The primary outcome of the clinical trial is labour market participation, defined as a dichotomized outcome, employment vs. on social transfer payment 12 months after hospital discharge.

SECONDARY OUTCOMES:
Return-to-work - Multi-state models of patients change in states from baseline to 12-months after hospital discharge | 12-months after hospital discharge
  3 multi-state models (working full-time, Working part-time, sick leave and the absorbing stated retired). Patients are not very likely to die during follow-up; this state may be superfluous. In the model working hours and retirement to private pensions will need to be assessed using self-reported data.
PRO: Readiness for return-to-work (RRTW) | 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  Readiness for return-to-work (RRTW) consisting of 22 items.
PRO: Degree of return-to-work | 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  Single items covering degree of RTW in hours weekly (compared to prior to the cardiac arrest), job describtion (changed Y/N) and job modification (changes Y/N).
PROM: EQ-5D-5L | Baseline (Hospital discharge), 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
PROM: Multidimensional fatigue inventory (MFI-20) | Baseline (Hospital discharge), 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  The MFI is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue.
PROM: The Hospital Anxiety and Depression Scale (HADS) | Baseline (Hospital discharge), 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  The questionnaire comprises seven questions for anxiety and seven questions for depression
PROM: The Pittsburgh Sleep Quality Index (PSQI) | Baseline (Hospital discharge), 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score
The Health Literacy Questionnaire (HLQ) | 2 weeks, 26 weeks and 52 weeks after hospital discharge
  HLQ has nine scales that each measure an aspect of the multidimensional construct of health literacy.
PROM: Disease specific health-related quality of life (HeartQoL) | 2 weeks, 12 weeks, 26 weeks and 52 weeks after hospital discharge
  The HeartQoL questionnaire comprises 14-items forming a physical, emotional subscales and a global score,
The Impact of Event Scale - Revised (IES-R) | 12 weeks, 26 weeks and 52 weeks after hospital discharge
  The Impact of Event Scale - Revised (IES-R) measures syptoms related to post-traumatic stress disorder (PTSD) The IES-R has 22 questions, that comprises a total subjective stress scale and three subscales (Intrusion, Avoidance, Hyperarousal)

OTHER OUTCOMES:
Montreal Cogntive Assessment (MoCA) | Baseline (Hospital discharge)
  The MoCA is a cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment
Assessment of Motor and Process Skills (AMPS) | Baseline (Hospital discharge)
  Measures the quality of a person's ADL task performance
Neurocognitive testing: Trail Making Test (TMT) Parts A and B | 1 month after hospital discharge
  the ability to think, reason, and remember
Neurocognitive testing: The Wechsler Adult Intelligence Scale | 1 month after hospital discharge
  WAIS-IV
Neurocognitive testing: The Repeatable Battery for the Assessment of Neuropsychological Status | 1 month after hospital discharge
  RBANS
Neurocognitive testing: Rey Complex Figure Test | 1 month after hospital discharge
  is a neuropsychological assessment in which examinees are asked to reproduce a complicated line drawing
Neurocognitive testing: The Symbol Digit Modalities Test (SDMT) | 1 month after hospital discharge
  A screening instrument to assess neurological dysfunction
Neurocognitive testing: The Five-Point Test | 1 month after hospital discharge
  The Five-Point Test is a test for measuring figural fluency functions
Neurocognitive testing: The Kohs Block test | 1 month after hospital discharge
  a performance test designed to be an IQ test
Neurocognitive testing: Animal fluency | 1 month after hospital discharge
  Verbal fluency tests are a kind of psychological test in which participants have to produce as many words as possible from a category in a given time
Neurocognitive testing: Fluency S-words | 1 month after hospital discharge
  Verbal fluency tests are a kind of psychological test in which participants have to produce as many words as possible from a category in a given time

CONTACTS AND LOCATIONS:
Overall Officials: Jan Christensen, PhD, Principal Investigator — Department of Occupational Therapy and Physiotherapy, Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
By contacting the corresponding author and upon reasonable request, de-identified data can be made available for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of all studies explicit stated in the Statistical Analysis Plan (SAP)
Access Criteria: By contacting the corresponding author and upon reasonable request, de-identified data can be made available for individual participant data meta-analysis.

REFERENCES:
- [Derived] Christensen J, Winkel BG, Kirkeskov L, Folke F, Winther-Jensen M, Eckhardt-Bentsen C, Kjaergaard J, Hassager C, Wagner MK. The ROCK trial-a multidisciplinary Rehabilitation intervention for sudden Out-of-hospital Cardiac arrest survivors focusing on return-to-worK: a pragmatic randomized controlled trial protocol. Trials. 2024 Feb 1;25(1):99. doi: 10.1186/s13063-024-07911-6. PMID 38303019
- See also: Related Info — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-024-07911-6